CLINICAL TRIAL: NCT01953627
Title: Laparoscopic Gynecologic Surgery With Robotic Assistance System Kymerax® : Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A00757-36; 2012-21 (Other: AP HM)
Record Dates: First submitted 2012-09-24; First posted 2013-10-01 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Gynecological Surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical procedure with the system Kymerax (Experimental)
  Interventions: Procedure: Surgical procedure with the system Kymerax; Device: The system Kymerax

INTERVENTIONS:
Procedure: Surgical procedure with the system Kymerax
Device: The system Kymerax

SUMMARY:
Laparoscopic robotic surgery (LSM) seems to increase quality of surgery. Diffusion of LSM is limited by cots of the only available system today. Kymerax® is a cheaper new system of LSM.

Aim : To evaluate feasibility of laparoscopy with Kymerax® system in different laparoscopic procedures in gynecology.

Material and methods : Observational study. Inclusion criteria were : patient requiring laparoscopic procedure in gynecology who give informed consent. The investigators evaluate procedures routinely performed by laparoscopy in gynecology.

Hypothesis : Procedures performed routinely in gynecology were feasible with Kymerax® system.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a following surgical procedure realized usually by coelioscopy:

Total hysterectomy or inter annexielle for mild or neoplastic pathology Promontofixation for genital prolapse Annexectomie or ovarian kystectomie for ovarian pathology Pelvic or lombo-aortic cleaning out for uterine cancer Tubaire Salpingectomie for pathology Rectovaginale partition Exérèse hurts of endometriosis

Exclusion Criteria:

* Patient refusing to participate in the study
* Patient understanding French.
* Minor waits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
assessment of Kymerax systemerax | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille; aubert AGOSTINI, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France